CLINICAL TRIAL: NCT03185468
Title: Intervention of Advanced or Metastatic Urothelial Bladder Cancer by 4SCAR-T Cell Therapies
Brief Title: Intervention of Bladder Cancer by CAR-T
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shenzhen Geno-Immune Medical Institute (Other)
Responsible Party: Principal Investigator, Lung-Ji Chang, President, Shenzhen Geno-Immune Medical Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIMI-IRB-17004
Record Dates: First submitted 2017-06-10; First posted 2017-06-14 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Bladder Cancer; Urothelial Carcinoma Bladder
Keywords: CAR T; Bladder
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 4SCAR-PSMA (Experimental): 4SCAR PSMA-modified T cells can recognize and kill tumor cells through the recognize of PSMA .This study will evaluate the side effects and effective doses of 4SCAR-PSMA T cells in treating refractory and recurrent solid tumors.
  Interventions: Genetic: 4SCAR-PSMA
- 4SCAR-FRa (Experimental): 4SCAR FRa-modified T cells can recognize and kill tumor cells through the recognize of FRa .This study will evaluate the side effects and effective doses of 4SCAR-FRa T cells in treating refractory and recurrent solid tumors.
  Interventions: Genetic: 4SCAR-FRa

INTERVENTIONS:
Genetic: 4SCAR-PSMA — PSMA-specific 4th Generation CART
  Arms: 4SCAR-PSMA
Genetic: 4SCAR-FRa — FRa-specific 4th Generation CART
  Arms: 4SCAR-FRa

SUMMARY:
This is a Phase I/II and multicenter study designed to evaluate the efficacy and safety of 4SCAR-T cells in participants with locally advanced or metastatic urothelial bladder cancer (UBC) who have no further treatment available.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically documented locally advanced or metastatic UBC (including renal pelvis, ureters, urinary bladder, and urethra)
2. Representative tumor specimens as specified by the protocol
3. Adequate hematologic and end organ function
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
5. Life expectancy greater than or equal to (>/=) 12 weeks
6. Measurable disease, as defined by RECIST v1.1

Exclusion Criteria:

1. Any approved anti-cancer therapy within 3 weeks prior to initiation of study treatment
2. Treatment with any other investigational agent or participation in another clinical trial with therapeutic intent within 28 days prior to enrollment
3. Active or untreated central nervous system (CNS) metastases as determined by computed tomography (CT) or magnetic resonance imaging (MRI) evaluation during screening and prior radiographic assessments
4. Leptomeningeal disease
5. Malignancies other than UBC within 5 years prior to Cycle 1, Day 1
6. Pregnant and lactating women
7. Significant cardiovascular disease
8. Severe infections within 4 weeks prior to infusion
9. Major surgical procedure other than for diagnosis within 4 weeks
10. History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins; known hypersensitivity or allergy to biopharmaceuticals produced in Chinese hamster ovary cells or any component of the atezolizumab formulation
11. History of autoimmune disease
12. Prior allogeneic stem cell or solid organ transplant
13. History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan
14. Positive test for human immunodeficiency virus (HIV) and/or active hepatitis B or hepatitis C or tuberculosis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival rate after receiving 4SCART infusion | 1 year
  to determine the efficacy of 4SCAR T cells
Using CTCAE 4 standard to evaluate the level of adverse events after receiving 4SCART infusion | 3 months
  to evaluate the level of adverse events with CTCAE 4

SECONDARY OUTCOMES:
The expansion and persistence of 4SCAR T cells | 1 year
  The investigators will monitor the expansion and functional persistence of 4SCAR T cells in the peripheral blood of patients and the correlation with antitumor effects
Immune responses after infusions | 3 months
  assessment of cytokine profile

CONTACTS AND LOCATIONS:
Overall Officials: Lung-Ji Chang, PhD, Principal Investigator — Shenzhen Geno-Immune Medical Institute
Locations (2):
- China (2):
  - Shenzhen Second People Hospital, Shenzhen, Gongdong
  - Shenzhen Geno-immune Medical Institute, Shenzhen, Guangdong

IPD SHARING:
Plan to Share IPD: No